CLINICAL TRIAL: NCT07303023
Title: Individualized Versus Standard Neck Prophylactic Irradiation in Nasopharyngeal Carcinoma: A Non-inferiority, Phase III, Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Individualized Neck Cervical Irradiation Prophylaxis Trial of NPC
Acronym: INCIPT-NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, MD. PhD., Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCIPT-NPC; 2507-83-01 (Registry Identifier: Shanghai Proton and Heavy Ion Center Institutional Review Board)
Record Dates: First submitted 2025-11-14; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: IMRT; carbon ion radiotherapy; Prophylactic Neck Irradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational arm (Experimental)
  Interventions: Radiation: Individualized Neck Irradiation
- control arm (Active Comparator): Standard Neck Irradiation
  Interventions: Radiation: Standard Neck Irradiation

INTERVENTIONS:
Radiation: Individualized Neck Irradiation — After confirmation of the radiotherapy technique, patients will be randomized. Patients in the investigational arm will receive bilateral upper neck irradiation covering at least Level II. If cervical lymph nodes are positive, the clinical target volume (CTV) will extend to 3 cm below the lowest level of metastatic (including suspected) lymph nodes.
  Arms: investigational arm
Radiation: Standard Neck Irradiation — Patients in the control arm will receive bilateral upper neck irradiation to level III; if upper neck nodes are positive, prophylactic irradiation of the lower neck will be performed.
  Arms: control arm

SUMMARY:
Based on the pattern of nasopharyngeal carcinoma cervical lymph node metastasis, which typically follows a sequential downward spread with rare skip metastases and a tendency for ipsilateral neck involvement, and in accordance with the latest international guidelines, we propose the following scientific hypothesis: individualized neck prophylactic irradiation for nasopharyngeal carcinoma based on the superior-to-inferior extent of metastatic lymph nodes is feasible. Specifically: if there is no lymph node metastasis, irradiation need only extend to the lower border of Level II; if there are suspected metastatic lymph nodes, a prophylactic dose of 55-60 Gy should be administered; the investigational arm will only require irradiation extending to 3 cm below the lowest level of metastatic (including suspected) lymph nodes in each neck.This study will prospectively enroll patients with N0-N3 stage nasopharyngeal carcinoma and randomize them to compare individualized neck irradiation based on the vertebral body level of metastatic lymph nodes versus selective upper neck prophylactic irradiation. The primary endpoint is neck recurrence-free survival. Secondary endpoints include overall survival, local recurrence-free survival and other survival data, incidence of acute and late neck radiation-induced injuries, and quality of life, aiming to validate the feasibility of individualized neck irradiation based on metastatic patterns.Photon IMRT and photon plus carbon-ion radiotherapy will serve as stratification factors, enabling further comparison of local control and toxicity between photon-carbon-ion therapy and photon-only (or proton) therapy. This study seeks to protect critical structures such as the thyroid, trachea, esophagus, and neck muscles while maintaining therapeutic efficacy, ultimately improving the quality of life for nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-inferiority, open-label, phase III randomized controlled clinical trial. A total of 462 patients will be enrolled, with an anticipated accrual period of three years and a follow-up period of three years post-enrollment.

Eligible patients will have newly diagnosed, non-metastatic nasopharyngeal carcinoma, staged as T1-4N0-3M0, Stage I-III according to the UICC/AJCC 9th edition staging system. After confirmation of the radiotherapy technique, patients will be randomized. Patients in the investigational arm will receive bilateral upper neck irradiation covering at least Level II. If cervical lymph nodes are positive, the clinical target volume (CTV) will extend to 3 cm below the lowest level of metastatic (including suspected) lymph nodes. Patients in the control arm will receive bilateral upper neck irradiation; if upper neck nodes are positive, prophylactic irradiation of the lower neck will be performed. Primary tumor and nodal CTV delineation for both arms will adhere to the 2024 international contouring guidelines for nasopharyngeal carcinoma.

Photon IMRT alone or photon IMRT plus carbon-ion radiotherapy will serve as stratification factors. The prescribed doses for photon IMRT alone are as follows: GTVp and GTVn: 66-70.4 Gy in 30-33 fractions; high-risk CTV1: 60 Gy in 30-33 fractions; low-risk CTV2: 50 Gy in 30-33 fractions. For the combined photon IMRT and carbon-ion radiotherapy arm, the prescription doses are: Photon IMRT - GTVp and GTVn: 55 Gy in 25 fractions; high-risk CTV1: 55 Gy in 25 fractions; low-risk CTV2: 50 Gy in 25 fractions. Carbon-ion boost - GTVp and GTVn: 15-18 Gy (RBE) in 6 fractions.

If indicated, patients will receive induction chemotherapy with the GP regimen (Gemcitabine 1000 mg/m² on Day 1 and Day 8, plus Cisplatin 75 mg/m² divided over three days) for 2-3 cycles. Concurrent chemotherapy, if administered, will consist of Cisplatin 80 mg/m² divided over three days, given every 3 weeks for 2 cycles.

Tumor response will be assessed by EBV-DNA levels and MRI at the end of induction chemotherapy, at the end of concurrent chemoradiotherapy, and three months after treatment completion. Follow-up visits will be scheduled every three months for the first two years post-treatment. Subsequent follow-up will be conducted as per protocol. Quality of life questionnaires, as specified by the study, will be completed before treatment, after treatment completion, and during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years.
2. Pathologically confirmed WHO type I, II, or III nasopharyngeal carcinoma.
3. Staged as T1-4N0-3 M0, Stage I-III according to the UICC/AJCC 9th edition staging system.
4. Absence of distant metastasis confirmed by systemic FDG PET/CT (or whole-body bone scan plus chest CT and abdominal ultrasound).
5. Ability to undergo MRI examination.
6. Adequate major organ function meeting radiotherapy requirements:

   1. Hematopoietic function: Hemoglobin ≥9 g/L, Platelets ≥100×10⁹/L, WBC ≥3.5×10⁹/L, Neutrophils ≥2.0×10⁹/L.
   2. Liver function: ALT and AST < 2.5 × ULN, Bilirubin < 1.5 × ULN.
   3. Renal function: Creatinine clearance ≥50 mL/min or serum creatinine within normal range.
   4. Patients with clinical symptoms will be evaluated based on specific manifestations.
7. ECOG performance status 0-1; absence of severe comorbidities (e.g., severe pulmonary hypertension, cardiovascular disease, peripheral vascular disease, severe chronic heart disease) that may preclude radiotherapy. Cardiac function class 1-2 (NYHA classification).
8. Life expectancy ≥12 months.
9. Patients must be informed of the study details and provide written informed consent.

Exclusion Criteria:

1. Pathology not confirming WHO type I, II, or III nasopharyngeal carcinoma.
2. Distant metastasis identified clinically or radiologically before treatment, or presence of skip metastases in cervical lymph nodes.
3. Pregnancy (confirmed by serum or urine β-HCG test) or lactation.
4. Unwillingness to provide informed consent.
5. Prior radiotherapy to the head and neck region.
6. Comorbidities or other factors that may contraindicate photon or carbon-ion therapy.
7. Inability to comply with regular follow-up due to psychological, social, familial, or geographical reasons.
8. Known allergy to chemotherapeutic agents (e.g., cisplatin, docetaxel, gemcitabine) or contrast media used in the study's imaging examinations.
9. Contraindication to contrast-enhanced MRI.
10. Major organ dysfunction, or severe uncontrolled concurrent infection or medical illness (e.g., decompensated cardiac, pulmonary, renal, or hepatic failure).
11. History of immunodeficiency (positive HIV test), other acquired/congenital immunodeficiency disorders, or history of organ/allogeneic bone marrow transplantation.
12. History of other malignancies prior to enrollment (except for basal cell carcinoma of the skin).
13. History of substance or alcohol abuse.
14. Any other condition deemed by the investigator to potentially lead to study discontinuation, including co-morbidities (including psychiatric) requiring concomitant treatment, severely abnormal laboratory values, or familial/social factors compromising patient safety or data integrity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
neck recurrence-free survival. | 3-year neck recurrence-free survival.

SECONDARY OUTCOMES:
overall survival | 3-year
local recurrence-free survival | 3-years
Locoregional Recurrence-Free Survival | 3 years
Distant Metastasis-Free Survival | 3 years

OTHER OUTCOMES:
incidence of acute and late neck radiation-induced injuries | 3-year

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Eye, Ear, Nose and Throat Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Sichuan Cancer Hospital & Institute, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Shanghai Proton and Heavy Ion Center, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Result] Zhu GL, Zhang XM, Yang KB, Tang LL, Ma J. Metastatic patterns of level II-V cervical lymph nodes assessed per vertebral levels in nasopharyngeal carcinoma. Radiother Oncol. 2023 Feb;179:109447. doi: 10.1016/j.radonc.2022.109447. Epub 2022 Dec 19. PMID 36549338
- [Result] Liu Y, Han Y, Liu F, Hu D, Chen Z, Wang P, Li J, Qin J, Jin F, Li Y, Wang J, Yi J. Involved site radiation therapy in stage I-III nasopharyngeal carcinoma with limited lymph node burden (ISRT-NPC) or elective region irradiation: a study protocol for a multicenter non-inferiority randomized controlled phase III clinical trial. BMC Cancer. 2023 Aug 3;23(1):724. doi: 10.1186/s12885-023-11212-7. PMID 37537541
- [Result] Liu Y, Yan W, Hu C, Huang X, Wang K, Qu Y, Chen X, Wu R, Zhang Y, Zhang J, Luo J, Li Y, Wang J, Yi J. Optimizing Cervical Target Volume in Patients with Nasopharyngeal Cancer Based On Nodal Drainage Distance. Clin Cancer Res. 2024 May 1;30(9):1801-1810. doi: 10.1158/1078-0432.CCR-23-3274. PMID 38349999
- [Result] Wang L, Wu Z, He Q, Li Y, Wang S, Li F, Wang H, Li W, Han Y. Distribution of regional lymph nodes metastasis in 870 cases of nasopharyngeal carcinoma and the suggestions for individualized elective prophylactic neck irradiation with intensity-modulated radiotherapy. Cancer Med. 2024 Feb;13(3):e6723. doi: 10.1002/cam4.6723. Epub 2023 Dec 29. PMID 38156901
- [Result] Xie DH, Wu Z, Li WZ, Cheng WQ, Tao YL, Wang L, Lv SW, Lin FF, Cui NJ, Zhao C, Ma J, Huang SM, Lu TX, Han YQ, Su Y. Individualized clinical target volume delineation and efficacy analysis in unilateral nasopharyngeal carcinoma treated with intensity-modulated radiotherapy (IMRT): 10-year summary. J Cancer Res Clin Oncol. 2022 Aug;148(8):1931-1942. doi: 10.1007/s00432-022-03974-7. Epub 2022 Apr 29. PMID 35486182
- [Result] Wu Z, Qi B, Lin FF, Zhang L, He Q, Li FP, Wang H, Han YQ, Yin WJ. Characteristics of local extension based on tumor distribution in nasopharyngeal carcinoma and proposed clinical target volume delineation. Radiother Oncol. 2023 Jun;183:109595. doi: 10.1016/j.radonc.2023.109595. Epub 2023 Mar 3. PMID 36870606
- [Result] Tang LL, Chen L, Xu GQ, Zhang N, Huang CL, Li WF, Mao YP, Zhou GQ, Lei F, Chen LS, Huang SH, Chen L, Chen YP, Zhang Y, Liu X, Xu C, Zhao Y, Li JB, Liu N, Xie FY, Guo R, Sun Y, Ma J. Reduced-volume radiotherapy versus conventional-volume radiotherapy after induction chemotherapy in nasopharyngeal carcinoma: An open-label, noninferiority, multicenter, randomized phase 3 trial. CA Cancer J Clin. 2025 May-Jun;75(3):203-215. doi: 10.3322/caac.21881. Epub 2025 Feb 19. PMID 39970442
- [Result] Huang CL, Zhang N, Jiang W, Xie FY, Pei XQ, Huang SH, Wang XY, Mao YP, Li KP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Zhou GQ, Ma J, Sun Y, Chen L, Tang LL. Reduced-Volume Irradiation of Uninvolved Neck in Patients With Nasopharyngeal Cancer: Updated Results From an Open-Label, Noninferiority, Multicenter, Randomized Phase III Trial. J Clin Oncol. 2024 Jun 10;42(17):2021-2025. doi: 10.1200/JCO.23.02086. Epub 2024 Mar 20. PMID 38507662
- [Result] Lin SJ, Guo QJ, Liu Q, Ng WT, Ahn YC, AlHussain H, Chan AW, Chow J, Chua MLK, Corry J, Han F, Gregoire V, Harrington KJ, Hu CS, Jensen K, Langendijk JA, Le QT, Lee NY, Lee V, Lin JC, Ma J, Mendenhall WM, O'Sullivan B, Ozyar E, Rosenthal DI, Tao YG, Wang RS, Wee J, Xu ZY, Yi JL, Yom SS, Fan DM, Mai HQ, Pan JJ, Lee AWM. International Consensus Guideline on Delineation of the Clinical Target Volumes at Different Dose Levels for Nasopharyngeal Carcinoma (2024 Version). Int J Radiat Oncol Biol Phys. 2025 Oct 1;123(2):415-431. doi: 10.1016/j.ijrobp.2025.05.019. Epub 2025 May 24. PMID 40419028
- [Result] Pan JJ, Mai HQ, Ng WT, Hu CS, Li JG, Chen XZ, Chow JCH, Wong E, Lee V, Ma LY, Guo QJ, Liu Q, Liu LZ, Xu TT, Gong XC, Qiang MY, Au KH, Liu TC, Chiang CL, Xiao YP, Lin SJ, Chen YB, Guo SS, Wong CHL, Tang LQ, Xu ZY, Jia YZ, Peng WS, Hu LP, Lu TZ, Jiang F, Cao CN, Xu W, Ma J, Blanchard P, Williams M, Glastonbury CM, King AD, Patel SG, Seethala RR, Colevas AD, Fan DM, Chua MLK, Huang SH, O'Sullivan B, Lydiatt W, Lee AWM. Ninth Version of the AJCC and UICC Nasopharyngeal Cancer TNM Staging Classification. JAMA Oncol. 2024 Oct 10;10(12):1627-35. doi: 10.1001/jamaoncol.2024.4354. Online ahead of print. PMID 39388190
- [Result] Lee AW, Ng WT, Pan JJ, Chiang CL, Poh SS, Choi HC, Ahn YC, AlHussain H, Corry J, Grau C, Gregoire V, Harrington KJ, Hu CS, Kwong DL, Langendijk JA, Le QT, Lee NY, Lin JC, Lu TX, Mendenhall WM, O'Sullivan B, Ozyar E, Peters LJ, Rosenthal DI, Sanguineti G, Soong YL, Tao Y, Yom SS, Wee JT. International Guideline on Dose Prioritization and Acceptance Criteria in Radiation Therapy Planning for Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2019 Nov 1;105(3):567-580. doi: 10.1016/j.ijrobp.2019.06.2540. Epub 2019 Jul 2. PMID 31276776
- [Result] Lee AW, Ng WT, Pan JJ, Poh SS, Ahn YC, AlHussain H, Corry J, Grau C, Gregoire V, Harrington KJ, Hu CS, Kwong DL, Langendijk JA, Le QT, Lee NY, Lin JC, Lu TX, Mendenhall WM, O'Sullivan B, Ozyar E, Peters LJ, Rosenthal DI, Soong YL, Tao Y, Yom SS, Wee JT. International guideline for the delineation of the clinical target volumes (CTV) for nasopharyngeal carcinoma. Radiother Oncol. 2018 Jan;126(1):25-36. doi: 10.1016/j.radonc.2017.10.032. Epub 2017 Nov 15. PMID 29153464
- [Result] Tang LL, Chen YP, Chen CB, Chen MY, Chen NY, Chen XZ, Du XJ, Fang WF, Feng M, Gao J, Han F, He X, Hu CS, Hu DS, Hu GY, Jiang H, Jiang W, Jin F, Lang JY, Li JG, Lin SJ, Liu X, Liu QF, Ma L, Mai HQ, Qin JY, Shen LF, Sun Y, Wang PG, Wang RS, Wang RZ, Wang XS, Wang Y, Wu H, Xia YF, Xiao SW, Yang KY, Yi JL, Zhu XD, Ma J. The Chinese Society of Clinical Oncology (CSCO) clinical guidelines for the diagnosis and treatment of nasopharyngeal carcinoma. Cancer Commun (Lond). 2021 Nov;41(11):1195-1227. doi: 10.1002/cac2.12218. Epub 2021 Oct 26. PMID 34699681